CLINICAL TRIAL: NCT01400373
Title: PRINCESS - Prehospital Resuscitation Intra Nasal Cooling Effectiveness Survival Study
Brief Title: Prehospital Resuscitation Intra Nasal Cooling Effectiveness Survival Study
Acronym: PRINCESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Erasme University Hospital (Other); University Hospital Hradec Kralove (Other); CHU de Charleroi (Other); University Hospital, Lille (Other); Karolinska University Hospital (Other); BeneChill, Inc (Industry)
Responsible Party: Principal Investigator, Leif Svensson, Leif Svensson, MD, PhD. Associate Professor in Cardiology. Karolinska Institutet, Södersjukhuset., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRINCESS 2010/383-32; NCT01328847 (obsolete NCT alias)
Record Dates: First submitted 2010-09-09; First posted 2011-07-22 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: Hypothermia, induced; Intra-arrest cooling; Cardiac arrest; Prehospital emergency care; Emergency Medical Services
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypothermia; Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients in the control group standard advanced cardiac life support care. Patients that achieve return of spontaneous circulation will be treated with hypothermia according to current guidelines upon arrival at the intensive care unit.
- Intervention (Experimental): Intra-arrest trans-nasal cooling with RhinoChill will be initiated during advanced cardiac life support. In patients achieving return of spontaneous circulation, trans-nasal cooling will continue until systemic cooling is started at the intensive care unit.
  Interventions: Device: Prehospital intra-nasal cooling with RhinoChill

INTERVENTIONS:
Device: Prehospital intra-nasal cooling with RhinoChill — Patients in the intervention group will receive prehospital intra-nasal cooling with RhinoChill as soon as possible during the resuscitation (i.e. intra-arrest). Intra-nasal cooling will be ongoing until systemic hypothermia is started at the intensive care unit.
  Arms: Intervention

SUMMARY:
Promising result of intra-arrest cooling on neurological intact survival in cardiac arrest patients has recently been published in the PRINCE-study in Circulation 2010.

The main purpose of this study is to determine whether prehospital intra-nasal cooling initiated during resuscitation, in addition to systemic cooling at hospital, increases neurological intact survival measured as cerebral performance category score (CPC-score)at 90 days in witnessed cardiac arrests outside hospital.

DETAILED DESCRIPTION:
Background:

The RhinoChill Device is a non-invasive, portable cooling device through which rapid cooling is achieved via the trans-nasal delivery of an evaporative coolant into the nasopharynx. Animal studies suggest a life-saving benefit for intra-arrest cooling.

Results from a European multicenter randomized trial (PRINCE - Pre Rosc Intra Nasal Cooling Effectiveness), published in Circulation in August 2010, demonstrate that intra-arrest trans-nasal evaporative cooling can be used safely and effectively in prehospital cardiac arrest without interfering with advanced cardiac life support protocols.

The outcome results among patients admitted to hospital showed a trend towards improved survival to hospital discharge in the treatment group (43.8% versus 31.0, p=0.26). The difference in neurologically intact survival was 34.4% vs 21.4%). In the subgroup of patients where cardiopulmonary resuscitation (CPR) was started by Emergency Medical Services personnel within 10 minutes (78 % of total number of patients) the difference in total survival between the groups was (56.5 versus 29.4, p=0.03). Neurologically intact survival for the corresponding subgroup was 43.5% vs 17.6%. In the treatment group, time to tympanic temperature of 34º was reached 3 hours faster (102 min versus 291 min, p=0.03) and time to core temperature 2 hours faster (155 min versus 284 min, p=0.13).

This study is powered to detect clinically significant changes in neurologically intact survival at 90 days after cardiac arrest. An interim analysis for safety and futility will be performed by an external committee after the first 200 patients have provided endpoint data. Conditional power for meeting the primary endpoint will if needed, be computed at that time, and if the interim results do not correspond to the primary endpoint, termination of the study for futility will be considered. Early stopping for efficacy reasons will only be considered if major outcome differences are seen between the groups according to the Haybittle rule with a p-value ≤0,001.

Intention to treat and per protocol analyses will be performed for all randomized patients. No imputed values will be used for patients for whom data is not available.

Stratified analyses will be performed for patients whose first recorded rhythm is VF/VT versus those in whom the first recorded rhythm is PEA or asystole. Stratification analyses will be performed for subjects where CPR was initiated within 10 minutes by a first responder. Stratified analyses will also be performed for subjects in the treatment group where cooling was started within 15 minutes.

Besides the specific endpoints listed below, substudies will be made to assess the following specific endpoints:

* Prehospital trans-nasal cooling significantly improve the systolic left ventricular function measured as LVEF (performed be Echo).
* Prehospital trans-nasal cooling significantly reduce the infarction size and area at risk and increase the systolic left ventricular function measured as LVEF (ECHO and MRI)in patients with AMI as cause of the cardiac arrest.
* Prehospital trans-nasal cooling significantly reduce in-hospital MACE (Major Adverse Cardiac Events) (i.e. death, reinfarction, stroke, cardiogenic shock, pulmonary oedema, recurrent cardiac arrest and need for.IABP.during hospital stay)
* Prehospital trans-nasal cooling significantly reduces the proportion of patients with cardiogenic shock
* Prehospital trans-nasal cooling significantly reduce days in ventilator, days at ICU and length of stay at hospital among survivors.
* To perform a metaanalysis in regards to ROSC, early and late survival as a pooled analysis of PRINCE data and PRINCESS 200 patientdata.
* Prehospital trans-nasal cooling significantly reduces peak-value of biochemical markers in patients treated with RhinoChill with 25% (measured at 12, 24, 36, 48 and 72 hours).
* To assess the development of end tidal CO2 during resuscitation in patients cooled prehospital wit trans nasal cooling

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Collapse was witnessed (heard or seen)
* Do not have a pulse
* Are unresponsive to external stimuli

Exclusion Criteria:

* Age ≥80 years
* Have an etiology of cardiac arrest due to trauma, severe bleeding, drug overdose, cerebrovascular accident, drowning, smoke inhalation, electrocution, hanging
* Already hypothermic (e.g., avalanche victim; found in the snow)
* Have an obvious barrier to placing intra nasal catheters (e.g., intranasal obstruction)
* Do Not Attempt to Resuscitate (DNAR) orders
* Have a terminal disease
* Known or clinically apparent pregnancy
* Have a known coagulopathy (except therapeutically induced)
* Are known to have a need for supplemental oxygen
* Achieve ROSC prior to randomization
* Response time (call to arrival) of the ambulance > 15 minutes

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2010-07-06 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Neurologically intact survival (CPC-cerebral performance categories scale 1-2) | 90 days after cardiac arrest
  The Cerebral Performance Categories (CPC) are used to describe neurological outcome. A CPC of 1 or 2 is considered "neurologically intact."
  1. - Good cerebral performance: little to no deficit.
  2. - Moderate cerebral disability: capable of independent activities of daily life
  3. - Severe cerebral disability: conscious, but dependent on others for daily support
  4. - Coma or vegetative state
  5. - Death or brain death

SECONDARY OUTCOMES:
Total survival | 90 days
Proportion of patients achieving Return of Spontaneous Circulation (ROSC). | 1 hour
Time to target temperature of 32-34º Celsius | 8-10 hours
Admitted alive to hospital | 2-4 hours
  Proportion of patients that are admitted alive to hospital

CONTACTS AND LOCATIONS:
Locations (2):
- Department of Intensive Care, Erasme University Hospital, Brussels, Belgium
- Department of Cardiology, Karolinska Institutet, Södersjukhuset, Stockholm, Sweden

REFERENCES:
- [Background] Nordberg P, Taccone FS, Castren M, Truhlar A, Desruelles D, Forsberg S, Hollenberg J, Vincent JL, Svensoon L. Design of the PRINCESS trial: pre-hospital resuscitation intra-nasal cooling effectiveness survival study (PRINCESS). BMC Emerg Med. 2013 Nov 25;13:21. doi: 10.1186/1471-227X-13-21. PMID 24274342
- [Background] Castren M, Nordberg P, Svensson L, Taccone F, Vincent JL, Desruelles D, Eichwede F, Mols P, Schwab T, Vergnion M, Storm C, Pesenti A, Pachl J, Guerisse F, Elste T, Roessler M, Fritz H, Durnez P, Busch HJ, Inderbitzen B, Barbut D. Intra-arrest transnasal evaporative cooling: a randomized, prehospital, multicenter study (PRINCE: Pre-ROSC IntraNasal Cooling Effectiveness). Circulation. 2010 Aug 17;122(7):729-36. doi: 10.1161/CIRCULATIONAHA.109.931691. Epub 2010 Aug 2. PMID 20679548
- [Derived] Nordberg P, Taccone FS, Truhlar A, Forsberg S, Hollenberg J, Jonsson M, Cuny J, Goldstein P, Vermeersch N, Higuet A, Jimenes FC, Ortiz FR, Williams J, Desruelles D, Creteur J, Dillenbeck E, Busche C, Busch HJ, Ringh M, Konrad D, Peterson J, Vincent JL, Svensson L. Effect of Trans-Nasal Evaporative Intra-arrest Cooling on Functional Neurologic Outcome in Out-of-Hospital Cardiac Arrest: The PRINCESS Randomized Clinical Trial. JAMA. 2019 May 7;321(17):1677-1685. doi: 10.1001/jama.2019.4149. PMID 31063573